CLINICAL TRIAL: NCT03392649
Title: Tragus Stimulation to Prevent Atrial Fibrillation After Cardiac Surgery: The TraP-AF Study
Brief Title: Tragus Stimulation to Prevent Atrial Fibrillation After Cardiac Surgery
Acronym: TraP-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Parasym Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB17-1365
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Results first posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Postoperative Atrial Fibrillation; Tragus Stimulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Group (No Intervention): At the end of cardiac surgery, the Parasym alligator clip was placed on the subject's tragus, but the Parasym was not turned on and the subject did not receive any stimulation. The clip was switched to the other ear every 4 hours for a total of 48 hours.
- Stimulation Group (Experimental): At the end of cardiac surgery, the Parasym alligator clip was placed on the subject's tragus, and the subject received continuous stimulation for 48 hours. The clip was switched to the other ear every 4 hours.
  Interventions: Device: Parasym

INTERVENTIONS:
Device: Parasym — Tragus stimulation was done using the Parasym device.
  Arms: Stimulation Group

SUMMARY:
Patients undergoing cardiac surgery, specifically a coronary artery bypass graft and/or heart valve replacement surgery, are at a higher risk for post-procedure atrial fibrillation (AF). AF is a condition in which the upper chambers of the heart do not contract normally and results in an irregular heartbeat. Recent studies have shown that tragus stimulation decreases the likelihood of AF in animals and humans. It has also been shown to reduce inflammation which may be related to post-procedure AF. Tragus stimulation involves stimulating a part of the outer ear, called the tragus, by sending a microcurrent through a small alligator clip. It is believed that tragus stimulation can affect the nervous system, which may reduce heart rate and lead to prevention of AF. The purpose of this study is to determine whether tragus stimulation in subjects undergoing cardiac surgery will lead to shorter occurrences, or even prevention, of AF.

DETAILED DESCRIPTION:
This was a single-blind study where patients were randomized tragus stimulation versus sham procedure and remained blinded to their treatment allocation. Both treatment options utilized similar equipment, namely the use of alligator clips which will be placed on the tragus and earlobe of the right ear for patients.

Prior to cardiac surgery, the discomfort threshold of both left and right tragus stimulation was determined for all participating patients. Intermittent electrode signals, or microcurrents, were delivered at 20 Hz with100 µsec pulse width with variable microampere (mA) output. The discomfort threshold was defined as the stimulation intensity in mA at which point patients experience discomfort. The stimulation intensity used in the study was set below the sensation and discomfort threshold. The clip was placed on the patient's ear at the end of surgery. Stimulation then continued, one ear alternating with the other, every 4 hours for a total of 48 hours. If the patient showed any sign of discomfort from stimulation, the intensity of stimulation was reduced to a level at which signs of discomfort disappears.

Follow-up was performed with a 14-day event monitor at the time of discharge, as clinically indicated. Echocardiography were assessed prior to study initiation and when clinically available in follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age, <90 years of age
2. Estimated life expectancy of at least 1 year at the time of enrollment
3. History of sinus rhythm or paroxysmal atrial fibrillation

Exclusion Criteria:

1. Patients ≥90 years of age, <18 years
2. Patients with known prior history of persistent or permanent AF
3. Atrial Fibrillation occurrence within the last 24 hours of procedure
4. Urgent or Emergency cases
5. Pregnant patients
6. Patients undergoing the following cardiac procedures: heart transplant, pulmonary thromboendarterectomy, isolated aortic arch procedures, congenital hear disease, ventricular assist device insertion, extracorporeal membrane oxygenation insertion, and surgical AF ablation
7. Antiarrhythmics prior to surgery (Class I and Class III)
8. High degree atrioventricular block requiring temporary pacing
9. Prior maze procedure for the treatment of AF

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav A. Upadhyay, MD, Principal Investigator — University of Chicago; Roderick Tung, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the University of Chicago Medical Center
Groups:
- Stimulation Group: At the end of cardiac surgery, the Parasym alligator clip was placed on the subject's tragus, and the subject received continuous stimulation for 48 hours. The clip was switched to the other ear every 4 hours.
  Parasym: Tragus stimulation has been done using the Parasym device.
Period: Overall Study
Arm/Group | Stimulation Group | Sham Group
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Group: At the end of cardiac surgery, the Parasym alligator clip was placed on the subject's tragus, but the Parasym was not turned on, and the subject did not receive any stimulation. The clip was switched to the other ear every 4 hours for a total of 48 hours.
- Total: Total of all reporting groups
Arm/Group | Stimulation Group | Sham Group | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [62 to 74.25] | 65.0 [59 to 75] | 66.0 [61 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 28 | 34 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27 | 32 | 59
  Race: African American | 4 | 6 | 10
  Race: Others | 9 | 3 | 12
Height(cm) [Median (Inter-Quartile Range); unit: cm] | 172.7 [163.8 to 177.8] | 177.8 [170 to 182.9] | 173 [165.1 to 182.9]
Weight(kg) [Median (Inter-Quartile Range); unit: kg] | 79.4 [71.05 to 98.3] | 92.3 [75.6 to 105.2] | 83.5 [72.6 to 104.1]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.17 [24.95 to 32.3] | 28.75 [24.55 to 32.55] | 28.56 [24.61 to 32.55]
NYHA Class [Count of Participants; unit: Participants] — Heart failure condition were classified according to New York Heart Association (NYHA) functional classification system and based on clinical assessments at the time of enrollment. Lower NYHA class is associated with less symptomatic heart failure, i.e., Class I: no limitations in physical activity; Class II: Patients are comfortable at rest but ordinary physical activity results in symptoms; Class III: Less than ordinary physical activity result in symptoms; Class IV: unable to carry out any physical activity without discomfort.
  Participants
    Class I | 0 | 1 | 1
    Class II | 10 | 14 | 24
    Class III | 21 | 15 | 36
    No heart failure symptoms noted | 9 | 11 | 20
Diabetes Mellitus [Count of Participants; unit: Participants] | 14 | 11 | 25
Hypertension [Count of Participants; unit: Participants] | 32 | 29 | 61
History of stroke or transient ischemic attack [Count of Participants; unit: Participants] | 6 | 4 | 10
Peripheral arterial disease [Count of Participants; unit: Participants] | 6 | 7 | 13
Creatinine [Median (Inter-Quartile Range); unit: micromoles/L] | 1.1 [0.9 to 1.225] | 0.9 [0.8 to 1.1] | 1.0 [0.9 to 1.1]
Chronic kidney disease [Count of Participants; unit: Participants] | 12 | 6 | 18
End-stage renal disease [Count of Participants; unit: Participants] | 3 | 2 | 5
Beta-blocker [Count of Participants; unit: Participants] | 26 | 16 | 42
Calcium channel blocker [Count of Participants; unit: Participants] | 13 | 11 | 24
Angiotensin converting enzyme inhibition or receptor blockade [Count of Participants; unit: Participants] | 22 | 20 | 42
Aldosterone blockade [Count of Participants; unit: Participants] | 1 | 2 | 3
Digoxin [Count of Participants; unit: Participants] | 0 | 1 | 1
Totally-endoscopic coronary artery bypass (TECAB) [Count of Participants; unit: Participants] | 4 | 5 | 9
Coronary artery bypass graft surgery (CABG) [Count of Participants; unit: Participants] | 25 | 17 | 42

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Episode of Atrial Fibrillation (AF) >30 Seconds
Description: Time to the first episode of atrial fibrillation (AF) that was greater than 30 seconds in patients who had AF. This was assessed on the review of patient chart and inpatient telemetry.
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Sham Group: At the end of cardiac surgery, the Parasym alligator clip was placed on the subject's tragus, but the Parasym was not turned on and the subject did not receive any stimulation. The clip has been switched to the other ear every 4 hours for a total of 48 hours.
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
hours | 53.1 [39.8 to 77.3] | 52.2 [28.7 to 62.3]
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Participants Hospitalized for >5 Days
Description: Number of participants with an overall length of hospitalization greater than five days.
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
Participants | 25 | 22
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.34, Chi-squared

3. Secondary Outcome: Overall Atrial Fibrillation (AF) Burden
Description: The total number of hours of atrial fibrillation (AF) burden as an inpatient.
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
hours | 24.7 [7.6 to 50.6] | 27.3 [12 to 89.3]
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Rate Control Medications Used for AF
Description: Number of participants that the management of their postoperative atrial fibrillation (AF) utilized the use of rate-controlling medications such as beta-blockers, calcium-channel blockers, or the use of digoxin.
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
Participants | 17 | 12
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.09, Fisher Exact

5. Secondary Outcome: Number of Participants With Antiarrhythmic Used to Treat AF
Description: Number of participants that antiarrhythmic was use to treat atrial fibrillation (i.e., use of amiodarone)
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
Participants | 16 | 10
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.16, Fisher Exact

6. Secondary Outcome: Number of Participants With Inotropes Used for Blood Pressure Support During AF
Description: The number of participants who management of their postoperative atrial fibrillation (AF) required the use of inotropic vasoactive or pressor medications for blood pressure (BP) support
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
Participants | 4 | 2
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.67, Fisher Exact

7. Secondary Outcome: Number of Participants With Stroke or Transient Ischemic Attack (TIA)
Description: The number of participants who suffered from a cerebral vascular accident (CVA) or transient ischemic attacks (TIA) for any cause during hospitalization was recorded.
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
Participants | 1 | 1
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 1.0, Chi-squared

8. Secondary Outcome: All-cause Mortality
Description: Number of participants who suffered from mortality due to any cause during the inpatient period
Time Frame: From end of surgery to end of hospitalization, up to 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation Group | Sham Group
Number analyzed (Participants) | 40 | 41
Participants | 3 | 0
Statistical Analysis 1: Comparison: Stimulation Group vs Sham Group; Test type: Superiority; p = 0.12, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the end of the surgery to the end of hospitalization, up to 1 month.
Arm/Group | Stimulation Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 3/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/41
Other Adverse Events (participants affected / at risk) | 0/40 | 1/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stimulation Group (N=40) | Sham Group (N=41)
Stroke or Transient Ischemic Attack (TIA) (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation Group (N=40) | Sham Group (N=41)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Discomfort from device with skin redness was noted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03392649/Prot_SAP_000.pdf